CLINICAL TRIAL: NCT01444859
Title: Effect of Trenev Trio®/Healthy Trinity® in Otherwise Healthy Adults With Recurrent Gastrointestinal Symptoms: a Double-blind, Randomized, Placebo-controlled, Parallel Group Study
Brief Title: Trenev Trio®/Healthy Trinity® for Recurrent Gastrointestinal Symptoms
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sprim Advanced Life Sciences (Other)
Collaborators: The National Institute of Probiotics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 110725-SUS-NIP-GIS-RA
Record Dates: First submitted 2011-09-28; First posted 2011-10-03 (Estimated); Last update posted 2012-10-24 (Estimated); Status verified 2011-12

CONDITIONS: Recurrent Gastrointestinal Symptoms
MeSH Terms: interventions — Probiotics; Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo capsule (Placebo Comparator): 40 subjects allocated to daily placebo capsule for 10 weeks
  Interventions: Dietary Supplement: Placebo
- Trenev Trio®/Healthy Trinity® (Experimental): 80 subjects allocated to Trenev Trio®/Healthy Trinity® for 10 weeks
  Interventions: Dietary Supplement: Trenev Trio®/Healthy Trinity®

INTERVENTIONS:
Dietary Supplement: Trenev Trio®/Healthy Trinity® — Trenev Trio®/Healthy Trinity® (1 capsule, 2x/day for 10 weeks), which offers a daily dose of: a) Lactobacillus acidophilus NAS strain (10 billion CFU), b) Bifidobacterium bifidum Malyoth strain (40 billion CFU), and c) Lactobacillus delbrueckii subspecies bulgaricus LB-51 strain (10 billion CFU)
  Other Names: Probiotic; Active
  Arms: Trenev Trio®/Healthy Trinity®
Dietary Supplement: Placebo — Daily placebo for 10 weeks
  Other Names: Inactive; Control
  Arms: Placebo capsule

SUMMARY:
Clinical trial to compare safety and effectiveness of 10-week supplementation with Trenev Trio®/Healthy Trinity® vs. placebo in otherwise healthy subjects with recurrent gastrointestinal symptoms.

DETAILED DESCRIPTION:
This study is a double-blind, randomized, placebo-controlled, parallel group trial comparing the safety and effectiveness of supplementation with Trenev Trio®/Healthy Trinity® vs. placebo in otherwise healthy subjects with recurrent gastrointestinal symptoms. Subjects will be recruited and, following successful completion of a 2-week run-in period, will be randomized to Trenev Trio®/Healthy Trinity® or placebo and will consume their assigned study product daily for 10 weeks. The study endpoints of this trial include relief of overall gastrointestinal symptoms, acid indigestion, abdominal cramping, constipation, diarrhea, gas, and bloating as well as product safety over the 10-week supplementation period.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Body mass index between 18.5 through 39.9 kg/m2
3. At least three symptoms rated between 4 to 6 in severity (moderate to severe discomfort) on a 1 to 7 scale, one of which must be acid indigestion as determined by the "Reflux Syndrome" score
4. Self-reported "acid indigestion" symptoms (including pain/discomfort beneath the breastbone, bitter fluid in the mouth, or bloating/nausea after eating) at least 3 times per week over the previous 4 weeks
5. Agree to use contraception throughout study period, unless postmenopausal or surgically sterile (females only)
6. Able to understand and voluntarily consent to the study and understand it's nature and purpose including potential risks, and side effects

Exclusion Criteria:

1. Any GSRS symptom rated a 7 in severity (very severe discomfort) on a 1 to 7 scale
2. Diagnosed gastrointestinal disease/complication or functional bowel disorder (e.g. IBS, functional constipation, IBD, ulcer, etc.) based on physical examination or documented medical history that, in the investigator's opinion, may affect subject safety or confound the evaluation of the study endpoints
3. Any non-gastrointestinal disease/complication that, in the investigator's opinion, may affect subject safety or confound the evaluation of the study endpoints
4. Regular (>3 days per week) prescription medication use for any gastrointestinal disease/condition
5. Recent (<6 months) abdominal surgery for any reason
6. Immunodeficiency
7. Recent change in anti-psychotic medication within the previous 3 months
8. Systemic steroid use within the prior month, excluding regular use of asthma medication
9. Pregnant female or breastfeeding
10. Eating disorder
11. Recent (within 2 weeks) antibiotic administration
12. History of alcohol, drug, or medication abuse
13. Daily consumption of probiotics, fermented milk, and/or yogurt
14. Known allergies to any substance in the study product
15. Participation in another study with any investigational product within 30 days of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-02; Primary Completion 2012-08 (Actual); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Mean total Gastrointestinal Symptom Rating Scale (GSRS) score | 10 weeks
Gastrointestinal Quality of Life Index (GIQLI) total score | 10 weeks

SECONDARY OUTCOMES:
Gastrointestinal Symptom Rating Scale subscores | 10 weeks
Gas severity | 10 weeks
Bloating severity | 10 weeks
Acid indigestion severity | 10 weeks
Abdominal cramping severity | 10 weeks
Stool consistency (measured with Bristol Stool Form Scale) | 10 weeks
Stool frequency | 10 weeks
Concomitant medication use | 10 weeks
Adverse event frequency | 10 weeks
Adverse event severity | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Duane Wombolt, MD, Principal Investigator — Clinical Research Associates of Tidewater; Jeffrey Stewart, MD, Principal Investigator — Research Across America; Michael Sinitsa, MD, Principal Investigator — Research Across America; Helen Stacey, MD, Principal Investigator — Diablo Clinical Research; Lydie Hazan, MD, Principal Investigator — Axis Clinical Trials; JoAnn Hattner, MPH, RD, Principal Investigator — Sprim ALS
Locations (5):
- United States (5):
  - Axis Clinical Trials, Los Angeles, California
  - Sprim ALS, San Francisco, California
  - Research Across America, West Lawn, Pennsylvania
  - Research Across America, Carrollton, Texas
  - Clinical Research Associates of Tidewater, Norfolk, Virginia